CLINICAL TRIAL: NCT01255514
Title: Sequential High-dose Dexamethasone and Response Adopted PAD (Bortezomib, Adriamycin, Dexamethasone) or VAD (Vincristine, Adriamycin, Dexamethasone) Induction Chemotherapy Followed by High-dose Chemotherapy With Autologous Stem Cell Transplantation for Newly Diagnosed Multiple Myeloma; Multicenter Phase 2 Study
Brief Title: Sequential High-dose Dexamethasone and Response Adopted PAD or VAD Induction Chemotherapy Followed by High-dose Chemotherapy With Autologous Stem Cell Transplantation for Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0510
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAD (Experimental): VAD : high dose dexamethasone -> response(CR, PR)-> VAD chemotherapy(vincristine + doxorubicin + dexamethasone)-> PBSC -> aSCT
  Interventions: Drug: high dose dexamethsone
- PAD (Experimental): PAD : high dose dexamethasone -> response(MR,NC,PD)-> PAD chemotherapy(bortezomib + doxorubicin + dexamethasone)-> PBSC -> aSCT
  Interventions: Drug: high dose dexamethsone

INTERVENTIONS:
Drug: high dose dexamethsone — high dose dexamethasone : 40mg/day , D1-D4, D9-D12, IV or PO, repeat every 21days for 2cycles

SUMMARY:
Complete Response (CR) plus near CR rate of VAD (Vincristine, Adriamycin, Dexamethasone) induction chemotherapy followed by ASCT in patients with newly diagnosed MM was about 50% and CR plus near CR rate of PAD (Bortezomib, Adriamycin, Dexamethasone) induction chemotherapy followed by ASCT in patients with newly diagnosed MM was about 60%. If the CR with near CR rate of sequential high-dose dexamethasone and response adopted PAD or VAD induction chemotherapy followed by ASCT is more than 60%, this combination will be accepted as active regimen that may be worth for investigating in phase III trial. But, if the CR with near CR rate of this regimen is lower than 50%, this has not a merit than VAD induction chemotherapy.

Based upon the above assumption, this trial was designed by using Simon's optimal two-stage testing procedure. Assuming a target level of interest, p1=0.6, and a lower activity level, p0=0.5. Initially 61 patients will be accrued. If 33 or more CR + near CR rate were observed, the trial will be continued. Accrual will be planned to a total of 190 patients. If total 106 or more patients were assessed as CR with near CR, sequential high-dose dexamethasone and response adopted PAD or VAD induction chemotherapy regimen will be accepted as active regimen. This design provides probability 0.05 of accepting drugs worse than p0 and probability 0.20 of rejecting drugs better than p1. If we assume that drop-out rate is 10%, total accrual patient will be 210.

Patient characteristics and toxicity will be evaluated by descriptive methods. Progression free survival and overall survival (median value, 95% confidence interval) will be calculated by Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of multiple myeloma (MM)
* Symptomatic MM (multiple myeloma with related organ or tissue damage)
* Previously untreated
* Age 20-65 years
* Performance status: ECOG 0-2
* Patient has measurable disease, defined as follows: For secretory multiple myeloma, measurable disease is defined as any quantifiable serum M-protein value and, where applicable, urine light chain of ≥200 mg/24 hours.
* For oligo-secretory multiple myeloma, measurable disease is defined as quantifiable light chain paraprotein on serum free light chain assay.
* For non-secretory multiple myeloma, measurable disease is defined as presence of soft tissue plasmacytoma(s) as determined by clinical examination or radiographic examination such as CT scan and magnetic resonance imaging (MRI), etc.
* Cardiac ejection fraction ≥ 50 % as measured by MUGA or 2D ECHO without clinically significant abnormalities
* Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value, Bilirubin < 2 X upper normal value
* Adequate hematological function: Platelet count ≥ 75 x 109/L, hemoglobin ≥ 8 g/dL, (Prior RBC transfusion or recombinant human erythropoietin use is allowed), absolute neutrophil count (ANC) ≥ 1.0 x 109/L
* A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause.
* Informed consent

Exclusion Criteria:

* Systemic AL amyloidosis, smoldering multiple myeloma or MGUS
* Patient with plasma cell leukemia (> 20% plasma cells in the PB and an absolute plasma cell count of at least 2000/μL)
* Previous chemotherapy or radiotherapy for the treatment of MM
* Patient is known to be Human Immunodeficiency Virus (HIV) positive
* Patient has known clinically active Hepatitis B or C
* Previous renal transplantation
* Severe peripheral neuropathy (Grade 2 or higher as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0)
* Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions :

  i. Uncontrolled or severe cardiovascular disease, including myocardial infarction, within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis ii. History of significant neurological or psychiatric disorders including dementia or seizures iii. Active uncontrolled infection (viral, bacterial or fungal infection) iv. Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or its ingredients (i.e., hypersensitivity to compounds containing boron or mannitol)
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10-30 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
CR+near CR | right after ASCT
  Assess the complete response (CR) + near CR (Immunofixation-positive CR) rate after autologous peripheral blood stem cell transplantation (ASCT)

SECONDARY OUTCOMES:
response of PAD/VAD chemotherapy | right after ASCT
  Assess the overall response of PAD/VAD chemotherapy and after ASCT

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - National Cancer Center, Goyang
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gill Hospital, Incheon
  - Severance Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul